CLINICAL TRIAL: NCT06991660
Title: The Effect of Sleep Hygiene Education Given in Line With the Health Promotion Model on Sleep Quality and Menopausal Symptoms
Brief Title: The Effect of Sleep Hygiene Education Given in Line With the Health Promotion Model on Sleep Quality and Menopause Symptoms
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Elif Yıldırım, principal investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023/4984
Record Dates: First submitted 2025-05-02; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-02

CONDITIONS: Absence of Menstrual Bleeding for at Least 12 Consecutive Months; No Communication Difficulties; Using a Mobile Phone; Becoming Literate; Not Using Sleeping Pills; Not Taking Any Supplements to Sleep
Keywords: menopause symptoms; midwife; sleep hygiene education; sleep quality; health promotion model
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: First interview: This interview, which was held at the ASM, included meeting the women in the intervention group, applying the pre-test data, explaining the purpose of the training, and determining the training location (ASM, the participant's home, etc.).
  Second interview: One week after the first interview, at the appointed location (ASM and the participant's home), the "Sleep Hygiene Training" prepared according to the individual characteristics - experiences and behavior-specific cognitive processes and behavioral outputs that are the components of the SGM was carried out, the "Sleep Diary" was introduced, the "Sleep Hygiene Training Booklet" and the "Sleep Diary" were distributed.
  Third interview: One week after the second interview, the repeat training, which constitutes the second session of the training, was carried out.
  Fourth interview: Obtaining the post-test data 4 weeks after the second interview.
  The researcher reminded the participants about the sleep diary via text m
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group (Experimental): First interview: This interview, which was held at the ASM, included meeting the women in the intervention group, applying the pre-test data, explaining the purpose of the training, and determining the training location (ASM, the participant's home, etc.).
  Second interview: One week after the first interview, at the appointed location (ASM and the participant's home), the "Sleep Hygiene Training" prepared according to the individual characteristics - experiences and behavior-specific cognitive processes and behavioral outputs that are the components of the SGM was carried out, the "Sleep Diary" was introduced, the "Sleep Hygiene Training Booklet" and the "Sleep Diary" were distributed.
  Third interview: One week after the second interview, the repeat training, which constitutes the second session of the training, was carried out.
  Fourth interview: Obtaining the post-test data 4 weeks after the second interview.
  The researcher reminded the participants about the sleep diary via text
  Interventions: Behavioral: sleep hygiene education
- control group (No Intervention): A total of two interviews were conducted with women in the control group who were not given any intervention. In the first interview, pre-test data were obtained using the Personal Introduction Form, MSDS and PSQI. In the interview held 6 weeks after the first interview, post-test data were obtained using MSDS and PSQI. Each interview lasted an average of 15-20 minutes.

INTERVENTIONS:
Behavioral: sleep hygiene education — This study will be conducted to examine the effects of sleep hygiene training, which is given to women in menopause to eliminate sleep problems and menopause symptoms that they often experience, on sleep and menopause symptoms experienced by women.
  Arms: training group

SUMMARY:
Health promotion is defined as the behaviors that a person exhibits for a long-term and high-standard life. Health promotion creates a sense of health in the individual, which makes the person feel more energetic and happy. The health promotion model primarily aims to treat the disease in the person. If the individual does not have a disease, their health is further improved. Sleep is one of the basic needs required for a person to continue their life in a healthy way. Some behaviors of people affect the quality and order of sleep. Sleep hygiene is the daily activities performed to improve the quality of sleep during sleep. Sleep hygiene education aims to avoid personal behaviors that affect a healthy sleep order and to exhibit behaviors that will positively affect sleep. Menopause is defined as the permanent cessation of the menstrual cycle as a result of the ovaries losing their activity. Menopause is one of the important stages of a woman's life. Some physical and psychological changes begin to occur in women who lose their fertility and enter menopause. These changes are generally called menopausal symptoms. These symptoms are; menstrual irregularity, hot flashes, sleep disorders, tension and depression, etc. The research was planned as an experimental pre-test and post-test, and the data will be collected before and after the face-to-face training given by the researcher. The effects of sleep hygiene training given in line with the health promotion model on sleep have been investigated in the literature, but no study has been found examining the effects of sleep hygiene training given in line with the health promotion model on sleep hygiene and menopausal symptoms of women in menopause. Therefore, it is thought that the research will contribute to the literature. The results obtained as a result of the study regarding the effects of sleep hygiene training given on sleep hygiene and menopausal symptoms will be taken into consideration by midwives.

ELIGIBILITY:
Inclusion Criteria:

* Not having menstrual bleeding for at least 12 consecutive months
* Not having difficulty communicating
* Using a mobile phone
* Being literate
* Not using sleeping pills
* Not taking any supplements to sleep.

Exclusion Criteria:

* Menstrual bleeding during the research period
* The participant wants to talk about his/her research.

Ages: 45 Years to 59 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women
Enrollment: 70 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index | first day encountered
  It was developed by Buysse et al. (1989) to assess sleep quality. It was adapted to Turkish by Ağargün et al. in 1996. The PSQI assesses the quality of an individual's sleep in the last month. While the individual answers 19 of the 24 questions in the PSQI, 5 questions are expected to be answered by the spouse or a roommate. The last 5 questions are directed only to the individual's relative in terms of clinical aspects and are not included in the scoring. The last of the questions asked as self-report questions is whether the individual has a roommate or spouse; this question is not used in the evaluation of the PSQI. There are different factors related to sleep quality in the self-report questions. The 18 items included in the scoring are divided into groups as 7 component scores. Some of the components are shown with only one item, while the other results in the classification of several items. Each component in the questions is worth 0-3 points.
Menopausal Symptoms Assessment Scale | first day encountered
  MSDÖ, developed by Schneider and colleagues in German to determine the level of menopause experienced by women, was translated and adapted into Turkish by Gürkan in 2005. The Likert-type scale consists of a total of 11 items covering menopausal complaints. Each item has three sub-dimensions, with the options 0: none at all, 1: mild, 2: moderate, 3: severe and 4: very severe. These are;
  1. Somatic symptoms sub-dimension: items 1, 2, 3, 11
  2. Psychological symptoms sub-dimension: items 4, 5, 6, 7
  3. Urogenital symptoms sub-dimension: items 8, 9, 10. The total score of the scale is calculated according to the scores given to each item. The lowest score on the scale is 0, and the highest score is 44. A high total score calculated at the end of the scale indicates that the participant has many complaints and that their standard of living is negatively affected.

SECONDARY OUTCOMES:
pittsburg sleep index | up to 4 weeks after registration
  It was developed by Buysse et al. (1989) to assess sleep quality. It was adapted to Turkish by Ağargün et al. in 1996. The PSQI assesses the quality of an individual's sleep in the last month. While the individual answers 19 of the 24 questions in the PSQI, 5 questions are expected to be answered by the spouse or a roommate. The last 5 questions are directed only to the individual's relative in terms of clinical aspects and are not included in the scoring. The last of the questions asked as self-report questions is whether the individual has a roommate or spouse; this question is not used in the evaluation of the PSQI. There are different factors related to sleep quality in the self-report questions. The 18 items included in the scoring are divided into groups as 7 component scores. Some of the components are shown with only one item, while the other results in the classification of several items. Each component in the questions is worth 0-3 points.
Menopausal Symptoms Assessment Scale | up to 4 weeks after registration
  MSDÖ, developed by Schneider and colleagues in German to determine the level of menopause experienced by women, was translated and adapted into Turkish by Gürkan in 2005. The Likert-type scale consists of a total of 11 items covering menopausal complaints. Each item has three sub-dimensions, with the options 0: none at all, 1: mild, 2: moderate, 3: severe and 4: very severe. These are;
  1. Somatic symptoms sub-dimension: items 1, 2, 3, 11
  2. Psychological symptoms sub-dimension: items 4, 5, 6, 7
  3. Urogenital symptoms sub-dimension: items 8, 9, 10. The total score of the scale is calculated according to the scores given to each item. The lowest score on the scale is 0, and the highest score is 44. A high total score calculated at the end of the scale indicates that the participant has many complaints and that their standard of living is negatively affected.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all IPD underlying results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR